CLINICAL TRIAL: NCT07206940
Title: Study of the Benefits of Virtual Reality Headsets for Reducing Anxiety in Patients Treated for Pleural Effusion or Pneumothorax Using Small-bore Chest Drainage Tubes - eSEDATION
Brief Title: Study of the Benefits of Virtual Reality Headsets for Reducing Anxiety in Patients Treated for Pleural Effusion or Pneumothorax Using Small-bore Chest Drainage Tubes
Acronym: eSEDATION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-AOI-01
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pneumothorax; Pleural Effusion; Drainage of Liquor
Keywords: Pneumothorax; Pleural Effusion; Drainage; virtual reality; anxiety reduction
MeSH Terms: conditions — Pneumothorax; Pleural Effusion | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reality virtual (Experimental): Standard support with reality virtual headset
  Interventions: Device: Drainage with Headset Hypno VR
- Standard of care (No Intervention): Standard support without reality virtual headset

INTERVENTIONS:
Device: Drainage with Headset Hypno VR — Pleural effusion and pneumothorax will be drained with the patient wearing the virtual reality headset.
  Arms: Reality virtual

SUMMARY:
Pleural effusion and pneumothorax are common conditions encountered in pulmonology departments and may require chest drainage. However, the chest drainage procedure can cause anxiety in patients, leading to discomfort during the procedure. The use of virtual reality (VR) for anxiety reduction has shown promising results in various medical contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient requiring Sledinger thoracic drainage for pneumothorax or pleural effusion in the pulmonology department of Nice University Hospital;
* Patient affiliated with social security;
* Signature of informed consent.

Exclusion Criteria:

* Immediate emergency situations;
* Anxiolytic, antidepressant, or psychotropic treatment already in place;
* Cognitive, behavioral, or psychiatric disorders;
* Language barrier;
* History of chest drainage or chest surgery;
* Hearing disorders without hearing aids;
* Vision disorders without corrective lenses (lack of binocular vision, blindness);
* Psychotic patients or patients diagnosed with psychiatric disorders;
* History of epilepsy;
* Current migraine;
* Patients for whom three-dimensional films are contraindicated (pacemaker or defibrillator);
* No social security coverage;
* Patients under guardianship/curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pain and Effects of personalized virtual reality | 18 months
  Compare the effects of personalized virtual reality support, compared to standard support, on pain in patients undergoing chest drainage with numerical pain scale from 0 to 10.
Anxiety and Effects of personalized virtual reality | 18 months
  Compare the effects of personalized virtual reality support, compared to standard support, on anxiety in patients undergoing chest drainage with numerical anxiety scale from 0 to 10.

SECONDARY OUTCOMES:
Pain assessment with or without VR headset based on heart rate | 18 months
  Heart rate will be used to assess the patient's pain. A heart rate between 55 and 85 beats per minute is normal.
Pain assessment with or without VR headset based on respiratory rate | 18 months
  Respiratory rate will be used to assess the patient's pain. A respiratory rate of 12 to 20 cycles per minute is normal.
Patient satisfaction | 18 months
  The evaluation will be based on the following question asked to the patient: "Are you satisfied overall with how the procedure went?" Possible answers: Yes/No.
Satisfaction of the paramedical team | 18 months
  The evaluation will be based on the following question asked to the paramedical team: "Are you generally satisfied with how the intervention went?" Possible answers: Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Nelly BANSE, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU Nice - Hôpital Pasteur 2, Nice, Alpes-Maritimes, France